CLINICAL TRIAL: NCT02119182
Title: Transforming Research and Clinical Knowledge in Traumatic Brain Injury
Acronym: TRACK-TBI
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1U01NS086090-01 (NIH); 1U01NS086090-01 (NIH)
Record Dates: First submitted 2014-03-22; First posted 2014-04-21 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Biomarkers; Neuroimaging; Psychological Health; Comparative Effectiveness Research
MeSH Terms: conditions — Brain Injuries, Traumatic; Psychological Well-Being | interventions — Blood Specimen Collection; DNA; RNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum, DNA, and RNA will be collected at the time of injury. Plasma, Serum, and RNA will be collected at Day 3 and Day 5 if patient is in the hospital, and at 2 weeks and 6 months post-injury. Samples will be banked at -80 degrees Celsius.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Comprehensive Assessment with MRI: * In-Person Outcome Assessment at 2 weeks, 6 months, and 12 months.
  * Phone Outcome Assessment at 3 months.
  * 3T Magnetic Resonance Imaging (MRI) at 2 weeks and 6 months.
  * Blood Draw for Plasma, DNA, Serum, RNA at baseline, in hospital (if applicable), 2 weeks, and 6 months (DNA at baseline only).
  Interventions: Behavioral: In-Person Outcome Assessment; Procedure: 3T Magnetic Resonance Imaging (MRI); Procedure: Blood Draw for Plasma, DNA, Serum, RNA
- Comprehensive Assessment without MRI: * In-Person Outcome Assessment at 2 weeks, 6 months, and 12 months.
  * Phone Outcome Assessment at 3 months.
  * Blood Draw for Plasma, DNA, Serum, RNA at baseline, in hospital (if applicable), 2 weeks, and 6 months (DNA at baseline only).
  Interventions: Behavioral: In-Person Outcome Assessment; Procedure: 3T Magnetic Resonance Imaging (MRI); Procedure: Blood Draw for Plasma, DNA, Serum, RNA
- Brief Assessment: • Telephone outcome assessment at 2 weeks, 3 months, 6 months, and 12 months.
  Interventions: Behavioral: Phone Outcome Assessment

INTERVENTIONS:
Behavioral: In-Person Outcome Assessment — NIH Flexible Outcome Assessment Battery Framework Measures In-Person at 2 Weeks, 6 Months, and 12 Months, and by Phone at 3 Months.
  Groups: Comprehensive Assessment with MRI; Comprehensive Assessment without MRI
Behavioral: Phone Outcome Assessment — NIH Flexible Outcome Assessment Battery Framework Measures by Phone at 2 Weeks, 3 Months, 6 Months, and 12 Months.
  Groups: Brief Assessment
Procedure: 3T Magnetic Resonance Imaging (MRI) — 3T Research MRI at 2 weeks and 6 months.
  Groups: Comprehensive Assessment with MRI; Comprehensive Assessment without MRI
Procedure: Blood Draw for Plasma, DNA, Serum, RNA — Blood Draw for Plasma, DNA, Serum, RNA at baseline, in hospital (if applicable), 2 weeks, and 6 months (DNA at baseline only).
  Groups: Comprehensive Assessment with MRI; Comprehensive Assessment without MRI

SUMMARY:
The overall goal of Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI) study is to determine the relationships among the clinical, neuroimaging, cognitive, genetic and proteomic biomarker characteristics for the entire spectrum of TBI from concussion to coma. TRACK-TBI will validate biomarkers and outcome measures for clinical trials, advance diagnostic and prognostic models for TBI and improve clinical trial design. The Investigators are enrolling patients within 24 hours of injury who present to a TRACK-TBI site with a brain injury that meets ACRM criteria and receives a clinically indicated head CT.

DETAILED DESCRIPTION:
Effective treatment of traumatic brain injury (TBI) remains one of the greatest unmet needs in public health. After 3 decades of failed clinical trials, a new approach is needed. Our proposal, Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI), establishes a public-private partnership of experienced TBI investigators, and philanthropic and industry collaborators, who share a mission to accelerate TBI research. TRACK-TBI will create a large, high quality database that integrates clinical, imaging, proteomic, genomic, and outcome biomarkers to establish more precise methods for TBI diagnosis and prognosis, refine outcome assessment, and compare the effectiveness and costs of TBI care.

The Investigators hypothesize that this approach will permit investigators to better characterize and stratify patients, allow meaningful comparisons of treatments and outcomes, and improve the next generation of clinical trials. The Investigators have built on the TRACK-TBI Pilot study (NCT01565551) and our team's precompetitive collaboration, forged by participation in the TBI Common Data Elements project (TBI-CDE) and the International TBI Research Initiative (InTBIR). Having provided the index dataset for the Federal Interagency TBI Research database (FITBIR), the Investigators now propose the following Specific Aims:

Specific Aim 1. To create a widely accessible, comprehensive TBI Information Commons that integrates clinical, imaging, proteomic, genomic, and outcome biomarkers from subjects across the age and injury spectra, and provides analytic tools and resources to support TBI research. Multi- disciplinary teams across 11 sites will enroll 3000 subjects of all ages across the injury spectrum of concussion to coma. Utilizing TBI-CDEs, along with uniform standards for acquiring multi-site MRI data, the Investigators will expand the TRACK-TBI Pilot informatics platform, leveraging existing informatics tools to populate FITBIR, yielding a resource for current and future TBI research and international collaboration.

Specific Aim 2. To validate imaging, proteomic, and genetic biomarkers that will improve classification of TBI, permit appropriate selection and stratification of patients for clinical trials, and contribute to the development of a new taxonomy for TBI. The Investigators hypothesize that validated imaging, proteomic, and genetic biomarkers will permit improved patient classification, beyond traditional categories of mild, moderate and severe TBI.

Subaim 2.1. To establish prognostic imaging biomarkers for TBI based on patho-anatomic analysis of CT and MRI, as well as quantitative MR volumetrics, diffusion tensor imaging (DTI), and resting state functional MRI (R-fMRI).

Subaim 2.2. To identify blood-based biomarkers that will provide additional diagnostic and prognostic information with which to identify TBI phenotypes that can be targeted by specific therapies.

Subaim 2.3. To identify common polymorphisms in candidate genes associated with outcome after TBI, and to elucidate causal molecular mechanisms of injury, response, and repair.

Subaim 2.4. To construct a multidimensional TBI classification system incorporating data from multiple domains that will define homogeneous classes of patients suitable for clinical trial inclusion.

Specific Aim 3. To evaluate a flexible outcome assessment battery comprised of a broad range of TBI common data elements that enables assessment of multiple outcome domains across all phases of recovery and at all levels of TBI severity. When compared with the current gold standard, the Glasgow Outcome Scale Extended (GOSE), the Investigators hypothesize that a flexible and more discriminating outcome battery reflecting multiple functional domains will more precisely and efficiently capture outcomes across the course of recovery, at all levels of TBI severity.

Subaim 3.1. To improve the granularity and breadth of TBI outcomes using a flexible outcome assessment battery that enables basic neurocognitive assessment in subjects too impaired to undergo standard neuropsychological testing, and comprehensive assessment of cognition, functional status, mental health, social participation, and quality of life in those cognitively intact enough to provide valid results.

Subaim 3.2. To determine the efficiency of a flexible outcome assessment battery, as compared with the GOSE, in reducing sample sizes needed to detect differences between groups.

Subaim 3.3. To identify specific TBI phenotypes amenable to targeted interventions, by relating patient classification factors (Subaim 2.4) to different outcome factor scores (Subaim 3.1).

Specific Aim 4. To determine which tests, treatments, and services are effective and appropriate for which TBI patients, and use this evidence to recommend practices that offer the best value. The Investigators will use established comparative effectiveness research (CER) and health economics methods to evaluate the ability of each clinical practice to improve outcomes while containing costs.

Subaim 4.1. To identify patients currently admitted to an ICU who could be safely and effectively cared for in a floor bed or discharged home with outpatient management, and to estimate the health and economic impact of changing the management of these patients.

Subaim 4.2. To determine whether routine follow up improves TBI outcomes and minimizes their economic burden.

Subaim 4.3. To assess variability in management of patients taking antiplatelet agents at the time of TBI, and the effect of management on progression of intracranial hemorrhage, need for craniotomy, and outcome.

The Investigators expect that achievement of these Specific Aims will advance our understanding of TBI, improve clinical trial design, lead to more effective patient-specific treatments, and improve outcome after TBI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-100 (some sites also enrolling pediatric patients)
* Documented/verified TBI by ACRM Criteria
* Injury occurred within 24 hours of ED arrival
* Acute brain CT as part of clinical care
* Visual acuity and hearing adequate for outcomes testing
* Fluency in English (some sites also enrolling Spanish speakers)

Exclusion Criteria:

* Significant polytrauma that would interfere with follow-up and outcome assessment
* Prisoners or patients in custody
* Pregnancy in female subjects
* Patients on psychiatric hold (e.g. 5150, 5250)
* Major debilitating baseline mental health disorders (e.g. schizophrenia or bipolar disorder) that would interfere with the validity of outcome assessment due to TBI
* Major debilitating neurological disease (e.g. stroke, CVA, dementia, tumor) impairing baseline awareness, cognition, or validity of outcome assessment due to TBI
* Significant history of pre-existing conditions that would interfere with likelihood of follow-up and validity of outcome assessment due to TBI (e.g. major substance abuse, alcoholism, end-stage cancers, learning disabilities, developmental disorders)
* Contraindications for MR (for CA+MRI cohort)
* Low likelihood of follow-up (e.g. participant or family indicating low interest, residence in another state or country, homelessness or lack of reliable contacts)
* Current participant in an interventional trial (e.g. drug, device, behavioral)
* Non-English speakers as most outcome measures are normed in the English language.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Investigators will enroll patients presenting to the Emergency Department with a history of acute TBI within the last 24 hours (acute injury) as per American Congress of Rehabilitation Medicine (ACRM) Criteria, in which the patient has sustained a traumatically induced* physiological disruption of brain function, as manifested by ≥ one of the following:
  Any period of loss of consciousness Any loss of memory for events immediately before or after the accident Any alteration of mental state at the time of the accident (feeling dazed, disoriented, and/or confused) Focal neurologic deficits that may or may not be permanent
  *Traumatically induced includes the head being struck, the head striking an object, or the brain undergoing an acceleration/deceleration movement without direct external trauma to the head.
Sampling Method: Non-Probability Sample
Enrollment: 2996 (Actual)
Dates: Start 2014-03-02 (Actual); Primary Completion 2019-06-22 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale - Extended (GOS-E) | 6 Months
  The Glasgow Outcome Scale - Extended (GOS-E) is the current gold standard of outcome for TBI.

SECONDARY OUTCOMES:
3T Brain Structural and Functional Magnetic Resonance Imaging (MRI) | 2 Weeks
  * Sagittal 3D T1 MPRAGE/IR-SPGR
  * Sagittal 3D T2* GRE
  * Axial Diffusion Tensor Imaging (DTI)
  * Axial Resting State Functional MRI (fMRI)
  * Sagittal 3D T2-FLAIR
  * Sagittal 3D T2
Blood Specimen for Analysis of Biomarkers and Genetics | Baseline Visit (In-Hospital)
  * 6.0ml blood for plasma and DNA
  * 6.0ml blood for serum
  * 2.5ml blood for RNA
TRACK-TBI Flexible Outcome Assessment Battery Framework (Composite Measure) | 2 Weeks
  Abbreviated Battery
  * GOS-E
  * Confusion Assessment Protocol - Cognitive (CAP-COG)
  * Coma Recovery Scale Revised (CRS-R)
  Comprehensive Assessment Battery
  * GOS-E
  * Expanded Disability Rating Scale (E-DRS-PI)
  * Rey Auditory Verbal Learning Test (RAVLT)
  * Trail Making Test (TMT)
  * Wechsler Adult Intelligence Scale IV (WAIS)
  * Brief Test of Adult Cognition by Telephone (BTACT)
  * Rivermead Post-Concussion Symptoms Questionnaire
  * Pain Intensity and Interference Instruments (PROMIS-PAIN)
  * Insomnia Severity Index (ISI)
  * Quality of Life After Brain Injury Overall Scale (QOLIBRI-OS)
  * Mayo-Portland Adaptability Inventory - Participation (MPAI-PART)
  * Satisfaction with Life Scale (SWLS)
  * 12-Item Short Form Survey (SF-12)
  * Alcohol Use Disorders Identification Test 3-Item (AUDIT-C)
  * 3-Item Drug Use Interview
  * Post-Traumatic Stress Disorder Checklist 5 (PCL-5)
  * Brief Symptom Inventory 18 (BSI18)
  * Participant Health Questionnaire 9 (PHQ-9)
TRACK-TBI Flexible Outcome Assessment Battery Framework (Composite Measure) | 3 Months
  Abbreviated Battery
  * GOS-E
  * Confusion Assessment Protocol - Cognitive (CAP-COG)
  * Coma Recovery Scale Revised (CRS-R)
  Comprehensive Assessment Battery
  * GOS-E
  * Expanded Disability Rating Scale (E-DRS-PI)
  * Rey Auditory Verbal Learning Test (RAVLT)
  * Trail Making Test (TMT)
  * Wechsler Adult Intelligence Scale IV (WAIS)
  * Brief Test of Adult Cognition by Telephone (BTACT)
  * Rivermead Post-Concussion Symptoms Questionnaire
  * Pain Intensity and Interference Instruments (PROMIS-PAIN)
  * Insomnia Severity Index (ISI)
  * Quality of Life After Brain Injury Overall Scale (QOLIBRI-OS)
  * Mayo-Portland Adaptability Inventory - Participation (MPAI-PART)
  * Satisfaction with Life Scale (SWLS)
  * 12-Item Short Form Survey (SF-12)
  * Alcohol Use Disorders Identification Test 3-Item (AUDIT-C)
  * 3-Item Drug Use Interview
  * Post-Traumatic Stress Disorder Checklist 5 (PCL-5)
  * Brief Symptom Inventory 18 (BSI18)
  * Participant Health Questionnaire 9 (PHQ-9)
TRACK-TBI Flexible Outcome Assessment Battery Framework (Composite Measure) | 12 Months
  Abbreviated Battery
  * GOS-E
  * Confusion Assessment Protocol - Cognitive (CAP-COG)
  * Coma Recovery Scale Revised (CRS-R)
  Comprehensive Assessment Battery
  * GOS-E
  * Expanded Disability Rating Scale (E-DRS-PI)
  * Rey Auditory Verbal Learning Test (RAVLT)
  * Trail Making Test (TMT)
  * Wechsler Adult Intelligence Scale IV (WAIS)
  * Brief Test of Adult Cognition by Telephone (BTACT)
  * Rivermead Post-Concussion Symptoms Questionnaire
  * Pain Intensity and Interference Instruments (PROMIS-PAIN)
  * Insomnia Severity Index (ISI)
  * Quality of Life After Brain Injury Overall Scale (QOLIBRI-OS)
  * Mayo-Portland Adaptability Inventory - Participation (MPAI-PART)
  * Satisfaction with Life Scale (SWLS)
  * 12-Item Short Form Survey (SF-12)
  * Alcohol Use Disorders Identification Test 3-Item (AUDIT-C)
  * 3-Item Drug Use Interview
  * Post-Traumatic Stress Disorder Checklist 5 (PCL-5)
  * Brief Symptom Inventory 18 (BSI18)
  * Participant Health Questionnaire 9 (PHQ-9)
3T Brain Structural and Functional Magnetic Resonance Imaging (MRI) | 6 Months
  * Sagittal 3D T1 MPRAGE/IR-SPGR
  * Sagittal 3D T2* GRE
  * Axial Diffusion Tensor Imaging (DTI)
  * Axial Resting State Functional MRI (fMRI)
  * Sagittal 3D T2-FLAIR
  * Sagittal 3D T2
Blood Specimen for Analysis of Biomarkers and Genetics | 2 Weeks
  * 6.0ml blood for plasma
  * 6.0ml blood for serum
  * 2.5ml blood for RNA
Blood Specimen for Analysis of Biomarkers and Genetics | 6 Months
  * 6.0ml blood for plasma
  * 6.0ml blood for serum
  * 2.5ml blood for RNA
TRACK-TBI Flexible Outcome Assessment Battery Framework (Composite Measure) | 6 Months
  Abbreviated Battery
  * GOS-E
  * Confusion Assessment Protocol - Cognitive (CAP-COG)
  * Coma Recovery Scale Revised (CRS-R)
  Comprehensive Assessment Battery
  * GOS-E
  * Expanded Disability Rating Scale (E-DRS-PI)
  * Rey Auditory Verbal Learning Test (RAVLT)
  * Trail Making Test (TMT)
  * Wechsler Adult Intelligence Scale IV (WAIS)
  * Brief Test of Adult Cognition by Telephone (BTACT)
  * Rivermead Post-Concussion Symptoms Questionnaire
  * Pain Intensity and Interference Instruments (PROMIS-PAIN)
  * Insomnia Severity Index (ISI)
  * Quality of Life After Brain Injury Overall Scale (QOLIBRI-OS)
  * Mayo-Portland Adaptability Inventory - Participation (MPAI-PART)
  * Satisfaction with Life Scale (SWLS)
  * 12-Item Short Form Survey (SF-12)
  * Alcohol Use Disorders Identification Test 3-Item (AUDIT-C)
  * 3-Item Drug Use Interview
  * Post-Traumatic Stress Disorder Checklist 5 (PCL-5)
  * Brief Symptom Inventory 18 (BSI18)
  * Participant Health Questionnaire 9 (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey T. Manley, MD, PhD, Study Director — University of California, San Francisco; Claudia S. Robertson, MD, Study Director — Baylor College of Medicine; David O. Okonkwo, MD, PhD, Study Director — University of Pittsburgh Medical Center; Ramon Diaz-Arrastia, MD, PhD, Study Director — University of Pennsylvania; Nancy R. Temkin, PhD, Study Director — University of Washington; Pratik Mukherjee, MD, PhD, Study Director — University of California, San Francisco; Joseph T. Giacino, MD, PhD, Study Director — Harvard Medical School, Spaulding Rehabilitation Hospital; Ann-Christine Duhaime, MD, Principal Investigator — Harvard Medical School, Massachusetts General Hospital; Dana P. Goldman, PhD, Principal Investigator — University of Southern California; Arthur W. Toga, PhD, Principal Investigator — University of Southern California; Kevin Smith, MSIS, Principal Investigator — University of Michigan; Opeolu M. Adeoye, MD, Principal Investigator — University of Cincinnati; Neeraj Badjatia, MD, MS, Principal Investigator — University of Maryland, College Park; Randall M. Chesnut, MD, Principal Investigator — University of Washington; Gillian A. Hotz, PhD, Principal Investigator — University of Miami; Christopher J. Madden, MD, Principal Investigator — University of Texas; Randall E. Merchant, PhD, Principal Investigator — Virginia Commonwealth University; Alex B. Valadka, MD, Principal Investigator — Seton Healthcare Family; Andrew I. Maas, MD, PhD, Principal Investigator — Antwerp University Hospital, Edegem, Belgium; David K. Menon, MD, PhD, Principal Investigator — University of Cambridge, Cambridge, United Kingdom; Isabelle Gagnon, PhD, MS, Principal Investigator — McGill University; Murray B Stein, MD, MPH, Study Director — University of California, San Diego; Ryan S Kitagawa, MD, Principal Investigator — The University of Texas Health Science Center, Houston; David M Schnyer, PhD, Principal Investigator — University of Texas at Austin; Vincent Y Wang, MD, PhD, MBA, Principal Investigator — Dell Seton Medical Center; David W Wright, MD, FACEP, Principal Investigator — Emory University; Michael McCrea, PhD, ABPP, Principal Investigator — Medical College of Wisconsin; Gregory Hawryluk, MD, PhD, Principal Investigator — University of Utah; Richard B Rodgers, MD, FAANS, Principal Investigator — Indiana University; Uzma Samadani, MD, PhD, Principal Investigator — University of Minnesota/Hennepin County Medical Center; Mitchell Cohen, MD, Principal Investigator — Denver Health and Hospital Authority; Cindy Harrison-Felix, PhD, FACRM, Principal Investigator — University of Colorado, Denver/Craig Hospital; Roland Torres, MD, Principal Investigator — University of Miami
Locations (23):
- United States (23):
  - University of California, San Francisco, San Francisco, California
  - Denver Health and Hospitals Authority, Denver, Colorado
  - University of Colorado/Craig Hospital, Englewood, Colorado
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spaulding Rehabilitation Hospital, Charlestown, Massachusetts
  - University of Minnesota/Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania/Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Dell Seton Medical Center, Austin, Texas
  - University of Texas at Austin, Austin, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - TIRR Memorial Hermann, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yue JK, Kanter JH, Barber JK, Huang MC, van Essen TA, Elguindy MM, Foreman B, Korley FK, Belton PJ, Pisica D, Lee YM, Kitagawa RS, Vassar MJ, Sun X, Satris GG, Wong JC, Ferguson AR, Huie JR, Wang KKW, Deng H, Wang VY, Bodien YG, Taylor SR, Madhok DY, McCrea MA, Ngwenya LB, DiGiorgio AM, Tarapore PE, Stein MB, Puccio AM, Giacino JT, Diaz-Arrastia R, Lingsma HF, Mukherjee P, Yuh EL, Robertson CS, Menon DK, Maas AIR, Markowitz AJ, Jain S, Okonkwo DO, Temkin NR, Manley GT; TRACK-TBI Investigators. Clinical profile of patients with acute traumatic brain injury undergoing cranial surgery in the United States: report from the 18-centre TRACK-TBI cohort study. Lancet Reg Health Am. 2024 Oct 17;39:100915. doi: 10.1016/j.lana.2024.100915. eCollection 2024 Nov. PMID 39497836
- [Derived] Yue JK, Etemad LL, Elguindy MM, van Essen TA, Belton PJ, Nelson LD, McCrea MA, Vreeburg RJG, Gotthardt CJ, Tracey JX, Coskun BC, Krishnan N, Halabi C, Eagle SR, Korley FK, Robertson CS, Duhaime AC, Satris GG, Tarapore PE, Huang MC, Madhok DY, Giacino JT, Mukherjee P, Yuh EL, Valadka AB, Puccio AM, Okonkwo DO, Sun X, Jain S, Manley GT, DiGiorgio AM; TRACK-TBI Investigators; Badjatia N, Barber J, Bodien YG, Fabian B, Ferguson AR, Foreman B, Gardner RC, Gopinath S, Grandhi R, Russell Huie J, Dirk Keene C, Lingsma HF, MacDonald CL, Markowitz AJ, Merchant R, Ngwenya LB, Rodgers RB, Schneider ALC, Schnyer DM, Taylor SR, Temkin NR, Torres-Espin A, Vassar MJ, Wang KKW, Wong JC, Zafonte RD. Prior traumatic brain injury is a risk factor for in-hospital mortality in moderate to severe traumatic brain injury: a TRACK-TBI cohort study. Trauma Surg Acute Care Open. 2024 Jul 24;9(1):e001501. doi: 10.1136/tsaco-2024-001501. eCollection 2024. PMID 39081460
- [Derived] Korley FK, Jain S, Sun X, Puccio AM, Yue JK, Gardner RC, Wang KKW, Okonkwo DO, Yuh EL, Mukherjee P, Nelson LD, Taylor SR, Markowitz AJ, Diaz-Arrastia R, Manley GT; TRACK-TBI Study Investigators. Prognostic value of day-of-injury plasma GFAP and UCH-L1 concentrations for predicting functional recovery after traumatic brain injury in patients from the US TRACK-TBI cohort: an observational cohort study. Lancet Neurol. 2022 Sep;21(9):803-813. doi: 10.1016/S1474-4422(22)00256-3. PMID 35963263
- [Derived] Galimberti S, Graziano F, Maas AIR, Isernia G, Lecky F, Jain S, Sun X, Gardner RC, Taylor SR, Markowitz AJ, Manley GT, Valsecchi MG, Bellelli G, Citerio G; CENTER-TBI and TRACK-TBI participants and investigators. Effect of frailty on 6-month outcome after traumatic brain injury: a multicentre cohort study with external validation. Lancet Neurol. 2022 Feb;21(2):153-162. doi: 10.1016/S1474-4422(21)00374-4. PMID 35065038
- [Derived] Campbell-Sills L, Jain S, Sun X, Fisher LB, Agtarap SD, Dikmen S, Nelson LD, Temkin N, McCrea M, Yuh E, Giacino JT, Manley GT; TRACK-TBI Investigators. Risk Factors for Suicidal Ideation Following Mild Traumatic Brain Injury: A TRACK-TBI Study. J Head Trauma Rehabil. 2021 Jan-Feb 01;36(1):E30-E39. doi: 10.1097/HTR.0000000000000602. PMID 32769835
- [Derived] Yue JK, Yuh EL, Korley FK, Winkler EA, Sun X, Puffer RC, Deng H, Choy W, Chandra A, Taylor SR, Ferguson AR, Huie JR, Rabinowitz M, Puccio AM, Mukherjee P, Vassar MJ, Wang KKW, Diaz-Arrastia R, Okonkwo DO, Jain S, Manley GT; TRACK-TBI Investigators. Association between plasma GFAP concentrations and MRI abnormalities in patients with CT-negative traumatic brain injury in the TRACK-TBI cohort: a prospective multicentre study. Lancet Neurol. 2019 Oct;18(10):953-961. doi: 10.1016/S1474-4422(19)30282-0. Epub 2019 Aug 23. PMID 31451409
- See also: NINDS Common Data Elements — https://www.commondataelements.ninds.nih.gov/Traumatic%20Brain%20Injury